CLINICAL TRIAL: NCT05983965
Title: Phase I Study to Evaluate Safety and Tolerability of Tazemetostat in Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: Study of Tazemetostat in Lymphoid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lauren Shea, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300011353
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: T-cell Lymphoma
Keywords: T-cell Lymphoma; Leukemia; Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia; Lymphoma | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort A (Experimental): T-cell Lymphomas
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Treatment: On day 1 and day 15 of the first cycle, and day 1 of all following cycles, the subject will have office visit with physical exam, vital signs, and lab tests. The subject will take tazemetostat twice a day by mouth continuously as an outpatient. If continuing on the treatment for more than 6 cycles, visits change to every 3 months.

SUMMARY:
Tazemetostat is an oral EZH2 inhibitor which has been FDA approved for adult patients with relapsed or refractory (R/R) follicular lymphoma (FL) whose tumors are positive for an EZH2 mutation as detected by an FDA-approved test and who have received at least 2 prior systemic therapies, and for adult patients with R/R FL who have no satisfactory alternative treatment option. We propose a study to evaluate the safety of tazemetostat in relapsed / refractory peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion criteria

1. Histologically confirmed peripheral T-cell lymphomas (PTCL) with allowed subtypes listed below as per the revised World Health Organization 2022 classification [6]:

   PTCL subtypes allowed
   1. PTCL-not otherwise specified (NOS)
   2. Nodal T-follicular helper cell lymphoma - angioimmunoblastic type, follicular type, or NOS
   3. Anaplastic Large Cell Lymphoma (ALK+)
   4. Anaplastic Large Cell Lymphoma (ALK-)
   5. Enteropathy-associated T-cell lymphoma
   6. Monomorphic epitheliotropic intestinal T-cell lymphoma
   7. Hepatosplenic T-cell lymphoma
   8. Subcutaneous panniculitis-like T-cell lymphoma
   9. Adult T-cell leukemia / lymphoma - lymphomatous, acute, or unfavorable chronic subtypes
2. Patients must have relapsed or refractory disease.

   1. Relapsed disease is defined when a patient progressed (>3 months) after achieving CR with a previous treatment
   2. Refractory disease is defined when a patient failed to achieve a CR or PR after a previous treatment
3. Patients received at least 1 prior therapy for PTCL.
4. At least one bi-dimensionally measurable nodal lesion, defined as ≥ 1.5 cm in its longest dimension, or one bi-dimensionally measurable extranodal lesion, defined as ≥ 1.0 cm in its longest diameter on fluorodeoxyglucose (FDG) positron emission tomography (PET)/computed tomography (CT) scan as defined by response criteria for PTCL
5. Age ≥ 18.
6. Patients with Hepatitis C can be included if they have completed therapy for hepatitis C with undetectable viral load.
7. Patients with Hepatitis B can be included if they are on suppressive therapy for hepatitis B infection and with no detectable viral load.
8. Patients with HIV can be included if they are on appropriate antiretroviral therapy, there is no interaction with the study drug, a CD4+ T-cell counts ≥ 350 cells/µL and no detectable viral load.
9. Adequate organ function as defined below unless attributed to disease involvement (Note: transfusions and growth factors allowed during screening; however, transfusion-dependency defined as requiring blood products ≥once per week not allowed):

   i. Liver function: No more than moderate hepatic impairment per NCI ODWG criteria - Total bilirubin ≤ 3X upper limit of normal (ULN), AST ≤ ULN (unless attributed to fatty liver or disease involvement).

   ii. Kidney function: CrCl > 30ml/min using Cockroft-Gault, based on actual weight.

   iii. ANC ≥ 1,000/µL, Platelet Count ≥ 75,000/ µL, Hemoglobin ≥ 8.0 g/dl.
10. Left ventricular ejection fraction (LVEF) defined by multiple-gated acquisition (MUGA) scan or echocardiogram within the institutional limits of normal.
11. Eastern Cooperative Oncology Group Performance Status of 0, 1, or 2.
12. A negative urine or serum pregnancy test is required for all women of childbearing potential within 1 week prior to enrolling on this trial and within 3 days of first dose of study drug. Note: Urine pregnancy tests that cannot be confirmed as negative require a confirmatory negative serum pregnancy test.

    Non-childbearing potential is defined as:
    * Postmenopausal: Defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, FSH measurements indicating post-menopausal status must be documented in patient's medical history.
    * Permanently sterile: Documented permanent sterilization e.g., hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
13. If female of childbearing potential, subject must not be pregnant or be breastfeeding and is required to have a negative urine or serum pregnancy test within 3 days prior to the first dose of study drug. In addition, females of childbearing potential must either practice complete abstinence or agree to use two effective methods of contraception simultaneously, beginning ≥ 28 days prior to start of tazemetostat, during tazemetostat treatment, and for at least 6 months after final dose of tazemetostat. See Appendix E regarding contraception guidelines.
14. Male subjects must either practice complete abstinence or agree to use a latex or synthetic condom during any sexual contact with a female of childbearing potential, from first dose of tazemetostat, during study treatment including dose interruptions, and for 3 months after last dose of tazemetostat. This applies even to males who have undergone successful vasectomy with medically confirmed azoospermia.
15. Willing and able to participate in all required evaluations and procedures in this study protocol including receiving intravenous administration of investigational product and being admitted, when required, for at least 24 hours during investigational product administration.

Exclusion criteria

1. Current evidence of central nervous system involvement.
2. Completion of an autologous hematopoietic stem cell transplantation within 3 months prior to first dose of study drug.
3. Prior allogeneic stem cell transplant within 6 months. The patient should not have any active GVH or should be on immune suppressive agents.
4. Completion of treatment with any radiotherapy, chemotherapy, antibody, immunoconjugates and/or another investigational drug ≤4 weeks (or 5 half-lives of the drug, whichever is shorter) prior to first dose of study drug. Patients may be enrolled after a minimum of 2 weeks of radiation if radiation was for palliative intent.
5. Prior therapy with an EZH2 inhibitor.
6. Inability to swallow and retain oral medications.
7. Pregnant women are excluded from this study.
8. Any active, concurrent, significant illness or disease (other underlying lymphoma) or clinically significant findings including psychiatric and behavioral problems, medical history and/or physical examination findings that would preclude the patient from participation in the study such as:

   i. Active infection requiring systemic therapy ≤10 days before the first dose of study drug; ii. Unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association [NYHA] II, III, IV;), myocardial infarction ≤6 months prior to first study drug, uncontrolled cardiac arrhythmia e.g., atrial fibrillation/flutter, cerebrovascular accidents ≤6 months before first dose of study drug; iii. Any severe or uncontrolled other disease or condition which might increase the risk associated with study participation.
9. Vaccination with live, attenuated vaccines within 28 days prior to the first dose of study medication.
10. Receiving systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents). The use of inhaled corticosteroids is permitted.
11. Corticosteroids ≥ 10 mg of prednisone within the last 7 days.
12. Has had a solid organ transplant within the last 3 years. Note: Patients who have had a solid organ transplant >3 years ago are eligible if there are no signs/symptoms of graft versus host disease (GvHD) and off immunosuppressive medications as per above.
13. Any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or myeloproliferative neoplasm (MPN).
14. Any prior history of T-cell lymphoblastic lymphoma (T-LBL)/T-cell acute lymphoblastic leukemia (T-ALL).
15. Patients with the following subtypes of lymphoma:

    i. T-cell prolymphocytic leukemia ii. T-large granular lymphocytic leukemia iii. NK-large granular lymphocytic leukemia iv. Aggressive NK-cell leukemia v. Breast implant-associated anaplastic large-cell lymphoma
16. Any other malignancy known to be active, with the exception of i. Cervical carcinoma of Stage 1B or less ii. Non-invasive basal cell or squamous cell skin carcinoma iii. Non-invasive, superficial bladder cancer iv. Prostate cancer with a current PSA level < 0.1 ng/mL v. Any curable or localized cancer with a CR of > 2 years' duration.
17. Any malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of tazemetostat.
18. Major surgery within 4 weeks before the first dose of study intervention. Note: Minor surgery (eg, minor biopsy of extracranial site, central venous catheter placement, shunt revision) is permitted within 3 weeks prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Identify the recommended phase II dose of Tazemetostat | 28 days
  The measurement will be the occurrence of a dose limiting toxicity (DLT) in the first cycle (28 days) after treatment initiation from the start of cycle 1 day 1.
  Measurements will be graded on a Hematologic Toxicity scale from grades 1 through 4 with grade 4 being worst grade.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No